CLINICAL TRIAL: NCT00828516
Title: Using Acupuncture and Moxibustion to Promote Wellbeing and Improve Quality of Life for Patients With Upper Body Lymphoedema Secondary to Cancer Treatment
Brief Title: Using Traditional Acupuncture in the Management of Cancer Treatment Related Lymphoedema
Acronym: AMWELL-SL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East and North Hertfordshire NHS Trust (Other Government)
Collaborators: Mount Vernon Cancer Centre at Mount Vernon Hospital (Other); International Lymphoedema Framework (Unknown); Lymphoedema Support Network (Unknown); University of Exeter (Other)
Responsible Party: Principal Investigator, Beverley de Valois PhD LicAc FBAcC, Research Acupuncturist, East and North Hertfordshire NHS Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000632850; LJMC-AMWELL-SL (Other Grant/Funding Number: NIHR RISC PB-PG-0407-10086); EU-20903
Record Dates: First submitted 2009-01-23; First posted 2009-01-26 (Estimated); Results first posted 2013-01-17 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2012-12

CONDITIONS: Breast Cancer; Head and Neck Cancer; Lymphedema
Keywords: lymphedema; male breast cancer; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; recurrent breast cancer; recurrent squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; stage I squamous cell carcinoma of the larynx; stage I verrucous carcinoma of the larynx; stage II squamous cell carcinoma of the larynx; stage II verrucous carcinoma of the larynx; recurrent adenoid cystic carcinoma of the oral cavity; recurrent mucoepidermoid carcinoma of the oral cavity; recurrent verrucous carcinoma of the oral cavity; stage I adenoid cystic carcinoma of the oral cavity; stage I mucoepidermoid carcinoma of the oral cavity; stage I verrucous carcinoma of the oral cavity; stage II adenoid cystic carcinoma of the oral cavity; stage II mucoepidermoid carcinoma of the oral cavity; stage II verrucous carcinoma of the oral cavity; stage I squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the lip and oral cavity; recurrent basal cell carcinoma of the lip; recurrent squamous cell carcinoma of the lip and oral cavity; stage I basal cell carcinoma of the lip; stage II basal cell carcinoma of the lip; recurrent metastatic squamous neck cancer with occult primary; recurrent lymphoepithelioma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; stage I lymphoepithelioma of the nasopharynx; stage I squamous cell carcinoma of the nasopharynx; stage II lymphoepithelioma of the nasopharynx; stage II squamous cell carcinoma of the nasopharynx; recurrent lymphoepithelioma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage I lymphoepithelioma of the oropharynx; stage I squamous cell carcinoma of the oropharynx; stage II lymphoepithelioma of the oropharynx; stage II squamous cell carcinoma of the oropharynx; recurrent esthesioneuroblastoma of the paranasal sinus and nasal cavity; recurrent inverted papilloma of the paranasal sinus and nasal cavity; recurrent midline lethal granuloma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; stage I esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage I inverted papilloma of the paranasal sinus and nasal cavity; stage I midline lethal granuloma of the paranasal sinus and nasal cavity; stage I squamous cell carcinoma of the paranasal sinus and nasal cavity; stage II esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage II inverted papilloma of the paranasal sinus and nasal cavity; stage II midline lethal granuloma of the paranasal sinus and nasal cavity; stage II squamous cell carcinoma of the paranasal sinus and nasal cavity; low-grade salivary gland mucoepidermoid carcinoma; recurrent salivary gland cancer; salivary gland acinic cell tumor; salivary gland adenocarcinoma; salivary gland adenoid cystic carcinoma; salivary gland anaplastic carcinoma; salivary gland malignant mixed cell type tumor; salivary gland poorly differentiated carcinoma; salivary gland squamous cell carcinoma; stage I salivary gland cancer; stage II salivary gland cancer; tongue cancer
MeSH Terms: conditions — Breast Neoplasms; Head and Neck Neoplasms; Lymphedema; Breast Neoplasms, Male; Squamous Cell Carcinoma of Head and Neck; Esthesioneuroblastoma, Olfactory; Salivary Gland Neoplasms; Tongue Neoplasms | interventions — Acupuncture Therapy; Moxibustion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Usual treatment plus acupuncture (Experimental): Acupuncture and moxibustion, individualised according to participant priorities, delivered once weekly for 7 treatments (Series 1) followed by 6 treatments (Series 2) if participant wishes to continue treatment
  Interventions: Other: Acupuncture and moxibustion

INTERVENTIONS:
Other: Acupuncture and moxibustion — Acupuncture is a form of traditional east Asian medicine that uses needles inserted superficially under the skin to stimulate sites on the body known as acupuncture points. Traditional practice encompasses moxibustion, the application of heat (usually from the smouldering herb artemisia vulgaris or mugwort) to stimulate the points by warming them.

SUMMARY:
RATIONALE: Acupuncture and moxibustion may improve well-being and quality of life in patients with lymphedema caused by breast cancer or head, neck, and throat cancer.

PURPOSE: This clinical trial is studying how well acupuncture given together with moxibustion works in improving well-being and quality of life in patients with breast cancer or head, neck, and throat cancer who are undergoing standard treatment for lymphedema.

DETAILED DESCRIPTION:
OBJECTIVES:

* To test the acupuncture and moxibustion treatment strategies to obtain a first measure of response for the approach(es) used in patients with breast cancer or head, neck, and throat cancer undergoing standard treatment for secondary lymphedema.
* To assess whether this treatment is an acceptable intervention to cancer patients with secondary lymphedema and to their health care professionals.
* To disseminate the data to begin to build the evidence base for using this treatment in the management of lymphedema.

OUTLINE: Patients undergo acupuncture and moxibustion therapy once weekly for 7 treatment (Series 1). After completion of therapy, patients may choose to continue treatment for an additional 6 treatments (Series 2).

Patients complete a set of 4 questionnaires (i.e., sociodemographic, Short-Form-36, Positive and Negative Affect Scale (PANAS), and Measure Yourself Medical Outcome Profile (MYMOP)) at the first treatment and then periodically during study. Patients also complete a series of follow-up questionnaires designed to elicit feedback about their acupuncture experience.

After completion of study treatment, patients are followed at 1 and 3 months.

ELIGIBILITY:
INCLUSION CRITERIA:

* male or female patients with either breast or head and neck cancer
* diagnosis of mild to moderate uncomplicated lymphoedema
* age 18 or over
* under the care of the lymphoedema service for at leas:
* two months (head and neck cancer patients)
* three months (breast cancer patients)
* no active cancer disease
* at least 3 months since prior active cancer treatment (surgery, radiotherapy, chemotherapy, intravenous treatment)
* more than 6 months since prior acupuncture treatment
* concurrent adjuvant hormonal therapy allowed
* concurrent anti-depressant medication allowed provided there has been no change in prescription or dosing within the past 3 months and patient intends to remain on the medication for the duration of study treatment and follow-up
* Able to understand and communicate in English
* Able to travel to the Lynda Jackson Macmillan Centre for treatment
* Able to attend treatment once weekly for at least 7 consecutive weeks
* Able to complete outcome measures

EXCLUSION CRITERIA:

* bilateral breast cancer
* advanced cancer disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2008-04; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beverley de Valois, PhD LicAc, Principal Investigator — Lynda Jackson Macmillan Centre at Mount Vernon Hospital
Locations (1):
- Lynda Jackson Macmillan Centre at Mount Vernon Cancer Centre, Northwood, United Kingdom

REFERENCES:
- [Background] de Valois B and Peckham R (2011) Treating the person and not the disease: acupuncture in the management of cancer treatment-related lymphoedema. European Journal of Oriental Medicine, 6(6), 37-49.
- [Result] de Valois BA, Young TE, Melsome E. Assessing the feasibility of using acupuncture and moxibustion to improve quality of life for cancer survivors with upper body lymphoedema. Eur J Oncol Nurs. 2012 Jul;16(3):301-9. doi: 10.1016/j.ejon.2011.07.005. Epub 2011 Sep 13. PMID 21917515
- [Result] de Valois B, Young T, Melsome E (2011) Acupuncture in lymphoedema management: a feasibility study. Journal of Lymphoedema. 6(2) 20-31.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment: June 2008 though May 2009. Participants recruited via the Mount Vernon Hospital Lymphoedema Service.
Groups:
- Clinical Phase: Breast cancer and head and neck cancer patients with lymphoedema secondary to cancer treatment. Acupuncture and moxibustion, individualised according to participant priorities, delivered once weekly for 7 treatments (Series 1) followed by a further 6 treatments (Series 2) if participant wishes to continue treatment.
Period: Clinical Phase: Series 1
Arm/Group | Clinical Phase
Started | 35
Completed | 33
Not Completed | 2
Not completed — Withdrawal by Subject | 2
Period: Clinical Phase: Series 2
Arm/Group | Clinical Phase
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Clinical Phase: Breast cancer and head and neck cancer patients with lymphoedema secondary to cancer treatment
Arm/Group | Clinical Phase
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 57.5 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 5
Region of Enrollment [Number; unit: participants]
  United Kingdom | 35

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Patient-specified and Reported Symptoms on the Measure Yourself Medical Outcome Profile (MYMOP)
Description: MYMOP is a questionnaire widely used for evaluating interventions based on holistic and participative principles. It enables respondants to specify and measure the treatment outcomes that are important to them.
Time Frame: Before 7th acupuncture treatment
Population: All participants completing 6 acupuncture treatments were analysed
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Usual Care Plus Traditional Acupuncture: All participants were considered stable and were undergoing maintenance treatment for lymphoedema, and were receiving adjunctive acupuncture treatment to promote wellbeing and improve quality of life
Arm/Group | Usual Care Plus Traditional Acupuncture
Number analyzed (Participants) | 32
units on a scale | 1.51 (0.96)
Statistical Analysis 1: Comparison: Usual Care Plus Traditional Acupuncture; There will be no improvement in MYMOP profile score after 6 acupuncture treatments; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — This was not adjusted for multiple comparisons; Mean Difference (Final Values) = 1.51, Standard Deviation 0.96 — MYMOP uses a 7-point scale, from 0 to 6, with "0" as good as it can be, and "6" as bad as it can be. Higher values represent a worse outcome

2. Primary Outcome: Change From Baseline in Patient-specified and Reported Symptoms on the Measure Yourself Medical Outcome Profile
Description: as for outcome 1
Time Frame: Before the 13th acupuncture treatment
Population: This was the number of participants who continued to, and completed, Series 2 of the treatments
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care Plus Traditional Acupuncture
Number analyzed (Participants) | 30
units on a scale | 1.32 (0.94)
Statistical Analysis 1: Comparison: Usual Care Plus Traditional Acupuncture; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — There will be no improvement in MYMOP profile score after 12 treatments; Mean Difference (Final Values) = 1.32, Standard Deviation 0.94 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Usual Care Plus Traditional Acupuncture
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No